CLINICAL TRIAL: NCT06184841
Title: Hepatic Arterial Infusion Chemotherapy Combined Sintilimab for Predominant Liver Metastasis From Esophageal Squamous Cell Carcinoma- A Pilot Study
Brief Title: HAIC Combined Sintilimab for Liver Metastasis From Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Guang Cao, Principal Investigator, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAIC FOR LMESC
Record Dates: First submitted 2023-01-03; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Arterial Infusion Chemotherapy; Liver Metastases; Esophageal Squamous Cell Carcinoma
Keywords: hepatic arterial infusion chemotherapy; liver metastasis; esophagus carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- esophageal squamous cell carcinoma with liver metastasis (Experimental): Patients with esophageal squamous cell carcinoma with liver metastasis have poor response to first-line treatment, especially those with advanced esophageal cancer with progression or recurrence in the liver.
  Interventions: Drug: HAIC combined with intravenous PD-1

INTERVENTIONS:
Drug: HAIC combined with intravenous PD-1 — Hepatic arterial chemoinfusion (HAIC) was used for interventional therapy with at least 2 cycles of hepatic arterial infusion. The intervention was started with sintilimab at the same time, 200mg each time, and the drug was repeated every 3 weeks.

SUMMARY:
Patients with liver metastasis from esophagus squamous (ESC) are usually offered systemic therapy. However, for those with predominant liver disease or failure of system therapy, local liver management becomes an option. This prospective single center study aimed to evaluate the efficacy and adverse events of hepatic arterial infusion chemotherapy (HAIC) using percutaneous catheter placement techniques for liver metastases from esophagus squamous (ESC).

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female, aged 18-75 years;
2. ECOG score 0-1;
3. Pathological diagnosis: metastatic esophageal squamous cell carcinoma confirmed by histological or cytological examination (excluding adenosquamous carcinoma mixed type and other pathological types).
4. Metachronous liver metastasis after esophagectomy, especially when liver was the only metastatic organ, or synchronous liver metastasis progressed after first-line medical treatment; Or liver metastasis is currently the main threat, and control of liver metastasis should be the main goal
5. predicted survival time ≥3 months.
6. Liver function: Child-Pugh score 5-7. ALT, AST, ALP< 2.5 times upper limit of normal, total bilirubin< 1.5 times upper limit of normal, PT, INR were < 1.5 times upper limit of normal, respectively. Bone marrow function was good (white blood cell ≥3.0 x 109/L, granulocyte ≥1.5 x 109/L, platelet ≥75 x 109/L, HGB≥100g/l), renal function was good (BUN < 40mg/dl, creatinine < 2mg/ml).
7. HBV infection, should have effective antiviral treatment, HBV DNA < 100IU/ml.
8. agree to be enrolled in the study, be willing to cooperate with the clinical research, and sign the informed consent.
9. Female subjects of childbearing age or male subjects whose sexual partner is a female of childbearing age should use effective contraception during the entire treatment period and for 6 months after the treatment period.

Exclusion Criteria:

1. age > 75 years old;
2. ECOG score ≥2;
3. poor liver function, Child-Pugh score > 7, or liver enzyme, coagulation, bilirubin and bone marrow function did not meet the inclusion criteria.
4. History of esophagogastric bleeding, hepatic encephalopathy, massive ascites, and abdominal infection.
5. lung, bone, mediastinal lymph nodes, multiple lower abdominal lymph nodes, pelvic lymph nodes and other distant metastases, unable to receive local radiotherapy.
6. The tumor was close to the intestinal tract and other organs, and it was difficult to tolerate interventional therapy; Patients with residual liver volume less than 800ml and difficult to tolerate interventional therapy.
7. allergic to Sintilimab.
8. patients had received previous immunotherapy, such as PD-1 antibody, PD-L1 antibody, CTLA4 antibody.
9. use of immunosuppressive drugs within the previous 4 weeks, excluding intranasal, inhaled, or other topical glucocorticoids or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/ day of prednisone or the equivalent dose of other glucocorticoids), and temporary use of glucocorticoids for the treatment of dyspnea in conditions such as asthma, chronic obstructive pulmonary disease, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 2 years
  Defined as the proportion of patients with Adverse events (AEs), Treatment Emergent Adverse events (TEAEs), Treatment-related AEs (TRAEs), immune-related AEs (irAEs), adverse events of special interest (AESI) and Serious Adverse events (SAE), assessed by NCI CTCAE v5.0

SECONDARY OUTCOMES:
The response rate of liver metastases | Up to 2 years
  Defined as proportion of patients who have a best response of CR or PR of liver metastases
The overall response rate ( ORR) | Up to 2 years
  Defined as proportion of patients who have a best response of CR or PR
The time to response (TTR) | Up to 2 years
  Defined as the time between the date of treatment start and objective tumor response
The duration of response (DOR) | Up to 2 years
  Defined as the time from first response (CR or PR) to the date of initial objectively documented progression or death due to any cause, whichever occurs first.
The progression free survival (PFS) | Up to 2 years
  Defined as the time from the date of treatment start to disease progression, or death due to any cause, whichever occurs first.
The overall survival (OS) | Up to 2 years
  Defined as the time from the date of treatment start to the date of death

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China